CLINICAL TRIAL: NCT05437536
Title: The Severe Von Willebrand Disease Patient Registry: a Longitudinal Natural History and Patient Outcomes Study
Brief Title: The Severe Von Willebrand Disease (sVWD) Patient Registry
Status: Recruiting | Type: Observational
Sponsor: VWD Connect Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: VWD-001
Record Dates: First submitted 2022-06-21; First posted 2022-06-29 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: VWD - Von Willebrand's Disease
Keywords: VWD; Severe VWD; VWD Type 1 Severe; VWD Type 1C; VWD Type 2A; VWD Type 2B Severe; VWD Type 2M Severe; VWD Type 2N Severe; VWD Type 3; Von Willebrand Disease; VWB; Von Willebrands Disease
MeSH Terms: conditions — von Willebrand Diseases; von Willebrand Disease, Type 3

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
A web-based registry will be created by the sponsor, VWD Connect Foundation (VCF), to collect data on patients with severe Von Willebrand Disease (sVWD). Data will be self-reported by patients and/or collected by registry personnel, as appropriate. The purpose of the sVWD Patient Registry is to create a database of well-characterized (with respect to demographics, medical history, symptoms, laboratory and genetic data, etc.) patients with sVWD for participation in retrospective and prospective research.

DETAILED DESCRIPTION:
A web-based registry will be created by the sponsor, VWD Connect Foundation (VCF), to collect data on patients with severe Von Willebrand Disease (sVWD). The initial launch of the registry will be limited to patients residing in the United States; however, the registry may be extended to other regions and countries upon the applicable regulatory approvals. Data will be self-reported by patients and/or collected by registry personnel, as appropriate. The purpose of the sVWD Patient Registry is to create a database of well-characterized (with respect to demographics, medical history, symptoms, laboratory and genetic data, etc.) patients with sVWD for participation in retrospective and prospective research. Patients who meet all eligibility criteria will be able to participate. Patients will be required to read and sign an Institutional Review Board (IRB)-approved informed consent form prior to any registry-specific activity taking place.

At the time of informed consent, participants will be asked to indicate if they are interested in being contacted by registry personnel for potential participation in future clinical trials and/or studies. Participants who opt out will not be contacted for future studies.

No clinical procedures, testing, or diagnostics will be required by virtue of registry participation. Participants will enter relevant data into a web-based registry portal at regular intervals.

Participants will be asked to complete questionnaires related to their sVWD (including diagnosis, symptoms, treatments, family history, quality of life, etc.) at the time of enrollment and at regular follow up intervals. Questionnaires will be released into the registry in phases as modules for participant completion. The first phase (ie, registry launch) will include, at minimum, modules on demographics, medical history, and concomitant medications. Additionally, the Self-Administered Bleeding Assessment Tool (Self-BAT) will be completed by participants at baseline and regular intervals. Questionnaire modules and the Self-BAT may also be administered in person by qualified registry personnel (e.g., at annual VCF conferences). Laboratory and genetic sequencing data will be provided by the participant, if available. Participants who have not completed a questionnaire in the registry website within a 12-month period will be contacted by registry personnel for follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Have a clinical diagnosis of Von Willebrand Disease (VWD) with any Von Willebrand factor level(s) < 20%
* Provide informed consent by participant or legally authorized representative
* Be willing and able to comply with study procedures and data collection
* Reside in the United States

NOTE: For inclusion criterion 1, it is not expected that participants will submit evidence of clinical diagnosis at screening; a participant's own confirmation that they have severe VWD will be sufficient for meeting the enrollment requirement and obtaining access to the registry. Laboratory values will be provided during the conduct of the study, and participants with Von Willebrand factor levels > 20% may be excluded from data analysis on a case-by-case basis in consultation with a subcommittee of the VWD Connect Foundation Medical and Scientific Advisory Board.

Exclusion Criteria:

* Have a clinical diagnosis of acquired VWD

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals diagnosed with severe VWD
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-12-10 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Outcomes are not applicable; this study is a patient registry. | At least 5 years
  Statistical analyses will focus on simple characterization of the registry.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Walsh, MD, PhD, Principal Investigator — Mt. Sinai School of Medicine; Mrinal Gounder, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Christina Morgenthaler, MS, MBA, Principal Investigator — VWD Connect Foundation
Locations (1):
- VWD Connect Foundation, Wellington, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified/coded data requests: The researcher will request the types of research or preparation for research that will be conducted with the data as part of the application process. After the VCF MSAB subcommittee approves the scientific/technical merit of the request, the registry research team will export and provide applicable de-identified data to the researcher. No information that would directly link the data to the participants will be included in the output data.